CLINICAL TRIAL: NCT06670768
Title: Myocardial Perfusion Quantification With Single Photon Emission Computed Tomography Using Multi-Pinhole Collimator Compared to Photon-Counting Coronary Computed Tomography Angiography
Brief Title: Myocardial Perfusion Quantification With SPECT Using Multi-Pinhole Collimator Compared to Photon-Counting Coronary CTA
Acronym: MY-FUSION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Prof. Maurovich-Horvat Pál, Head of Clinic for Medical Imaging, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OGYÉI/64876-6/2023
Record Dates: First submitted 2024-10-24; First posted 2024-11-01 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease; Coronary Computed Tomography Angiography; SPECT; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Myocardial Ischemia; Coronary Disease; Chest Pain
Keywords: Coronary Artery Disease,; Myocardial Perfusion Imaging; Myocardial Perfusion Imaging Absolute Quantification; Myocardial Flow Reserve; Plaque volume
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Myocardial Ischemia; Coronary Disease; Chest Pain

STUDY DESIGN:
Intervention Model Description: Consecutive patients with suspected coronary artery disease are enrolled. Patients are referred to dynamic and static MPI using 99mTc radionuclide imaged by SPECT, following coronary CTA examination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Consecutive patients with moderate pre-test probability according to CAD consortium (Experimental): Patients undergo dynamic and static MPI SPECT and cardiac CT within 30-days.
  Interventions: Diagnostic Test: Stress Dynamic MPI SPECT; Diagnostic Test: Stress Static MPI SPECT; Diagnostic Test: Rest Dynamic MPI SPECT; Diagnostic Test: Rest Static MPI SPECT; Diagnostic Test: Cardiac CT

INTERVENTIONS:
Diagnostic Test: Stress Dynamic MPI SPECT — BMI standardized radiopharmaceutical injection in pharmacological stress (dipyridamole or adenosine) is performed under the SPECT camera to record the temporal distribution of the activity. A one-day protocol and multi-pinhole collimator are used.
Diagnostic Test: Stress Static MPI SPECT — 30-60 minutes after stress dynamic SPECT imaging is performed, an ECG-gated static SPECT MPI is conducted with a conventional LEHR collimator.
Diagnostic Test: Rest Dynamic MPI SPECT — 3 hours after the stress phase, the rest phase is also recorded. A radiopharmaceutical injection with a three-fold dose at rest is performed under the SPECT camera to record the temporal distribution of the activity. A one-day protocol and multi-pinhole collimator are used.
Diagnostic Test: Rest Static MPI SPECT — 30-60 minutes after rest, dynamic SPECT imaging is performed, and an ECG-gated static SPECT MPI is conducted with a conventional LEHR collimator.
Diagnostic Test: Cardiac CT — Within 30 days of MPI SPECT imaging, a cardiac CT is performed for every patient, including a native calcium-scoring scan and a coronary CT angiography as a reference standard. A photon-counting detector CT is used.

SUMMARY:
This prospective study aims to compare functional abnormalities detected using myocardial perfusion SPECT imaging (MPI SPECT) with the extent and severity of anatomical findings on coronary computed tomography angiography (coronary CTA). Additionally, the investigators aim to enhance the diagnostic value of MPI SPECT by quantifying myocardial blood flow and utilizing myocardial flow reserve calculated from dynamic SPECT images.

50 patients with suspected coronary artery disease are anticipated to be enrolled. Pharmacological stress and rest-phase dynamic and static MPI SPECT following an additional coronary CTA scan are to be performed. The obtained multimodality imaging data (functional and anatomical parameters) are planned to be compared and subjected to statistical analysis. The results of this study are expected to improve risk assessment for patients with moderate cardiovascular risk and enhance the diagnostic performance of MPI SPECT.

DETAILED DESCRIPTION:
Diagnostic management of patients with moderate clinical likelihood of obstructive coronary artery disease (CAD) remains challenging. Myocardial perfusion SPECT imaging (MPI SPECT) is a widely available and cost-effective modality that provides functional information on segmental perfusion defects. However, conventional static MPI SPECT has moderate diagnostic performance in identifying subclinical coronary atherosclerosis.

The novel multi-pinhole (MPH) collimator technology with a three-detector SPECT camera (AnyScan® TRIO SPECT/CT, Mediso Ltd., Hungary) enables temporal and spatial resolution, absolute quantification of stress and rest myocardial blood flow (sMBF and rMBF), and calculated myocardial flow reserve (MFR), overcoming the difficulties of semi-quantitative evaluation.

This study aims to investigate the association between quantitative MFR, semi-quantitative functional parameters of dynamic, static MPI SPECT, and coronary CTA-based plaque metrics. Flow parameters of myocardial wall segments will be corresponded to the appropriate coronary artery based on the CT-assessed anatomy. Furthermore, the investigators aim to build statistical models representative of clinical scenarios to test the diagnostic accuracy of the MPH collimator.

In this prospective study, 50 patients with moderate cardiovascular pre-test probability (PTP) referred to either coronary CTA or MPI SPECT are anticipated to be enrolled. Cardiovascular PTP is estimated according to the CAD consortium based on age, sex, type of chest pain, and cardiovascular risk factors. Patients with a history of coronary artery bypass graft implantation, left or right bundle branch block, and atrial fibrillation will be excluded. Participants will be subjected (1) to dynamic and (2) static MPI SPECT (pharmacological stress and rest) and (3) to coronary CTA within 30 days. Patients undergoing pharmacological stress (dipyridamole or adenosine) dynamic MPI SPECT, which will be performed with AnyScan® TRIO SPECT/CT (Mediso Ltd.). Imaging will be started at the time of the radiopharmaceutical administration both in stress and rest, captured for 15 minutes in list mode. BMI-standardized doses of 99m-Tc will be used, with a same-day acquisition protocol, resulting in a three-fold increase for the rest phase compared to stress. Following each phase of dynamic acquisition in 30-60 minutes, an ECG-gated static MPI SPECT will be performed using a conventional LEHR collimator.

Data, such as sMBF, rMBF, MFR, summed stress score (SSS), summed rest score (SRS), summed difference score (SDS), as well as visually evaluated perfusion defect severity and extent will be determined from MPI SPECT. Within 30 days of MPI SPECT, coronary CTA with Calcium Score assessment will also be performed using a photon-counting detector CT (NAEOTON Alpha, Siemens Healthineers, Germany). Coronary CTA will be analyzed as follows: coronary artery calcium score (CACS), the severity of luminal stenosis, total plaque volume, quantitative plaque composition, and CT-derived fractional flow reserve (FFR). The following additional anamnestic covariants will be used: age, sex, and cardiovascular risk factors such as type of chest pain, diabetes mellitus, hypertension, smoking, obesity, and dyslipidemia.

The investigators hypothesized that dynamic MPI SPECT may prove to be superior to semi-quantitative static MPI SPECT in detecting CAD. Furthermore, MFR data combined with CACS may improve the diagnostic accuracy of MPI SPECT and guide the selection of patients for invasive coronary angiography.

MPI SPECT and coronary CTA data will be analyzed on-site at Semmelweis University, Hungary. The results will be available after the completion of patient enrollment.

ELIGIBILITY:
Inclusion Criteria:

* suspected coronary artery disease
* referred to coronary CTA or SPECT MPI by the patient's physician
* agrees to the other imaging modality that was not indicated by their physician (coronary CTA or SPECT MPI)
* suitable for informed consent

Exclusion Criteria:

* moderate or severe aortic valve stenosis
* atrial fibrillation
* pregnancy or breastfeeding
* history of coronary artery bypass graft implantation
* history of stent implantation
* chronic renal failure (eGFR < 30 ml/m2)
* active oncological treatment
* congenital heart disease
* left or right bundle branch block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
The association between Myocardial Flow Reserve (MFR) and total non-calcified plaque volume as assessed by coronary CTA. | As soon as all required data is available but not later than study completion, an avarage of one year.
  Predictive value of MFR on vessel and participant level, expressed as the ratio of Stress/Rest Myocardial Blood Flow (sMBF/rMBF). The total non-calcified plaque volume will be measured by PCD-CT.

SECONDARY OUTCOMES:
Predictive Value of Myocardial Flow Reserve (MFR) to CT-derived Fractional Flow Reserve (FFR-CT) | As soon as all required data is available but not later than study completion, an avarage of one year.
  The predictive value of MFR on vessel and participant levels is expressed as the ratio of stress/rest myocardial blood flow (sMBF/rMBF) to FFR-CT of 0.8 or less in any coronary artery. FFR-CT values are defined as follows: greater than 0.8 is normal, 0.76-0.8 is borderline, and 0.75 or less is abnormal.
Predictive Value of stress Myocardial Blood Flow (sMBF) to lumen stenosis extent on coronary CTA | As soon as all required data is available but not later than study completion, an avarage of one year.
  The predictive value of sMBF on vessel and participant level, derived from dynamic MPI SPECT, expressed in unit of ml/min/g to luminal stenosis extent. The severity of luminal stenosis is defined as follows: no stenosis, 1-24% minimal, 25-49% mild, 50-69% moderate, 70-99% severe, occlusion.
Predictive Value of stress Myocardial Blood Flow (sMBF) to CT-derived Fractional Flow Reserve (FFR-CT) | As soon as all required data is available but not later than study completion, an avarage of one year.
  The predictive value of sMBF on vessel and participant levels, derived from dynamic MPI SPECT, is expressed in a unit of ml/min/g to FFR-CT of 0.8 or less in any coronary artery. FFR-CT values are defined as follows: greater than 0.8 is normal, 0.76-0.8 is borderline, and 0.75 or less is abnormal.
Correlation of Myocardial Flow Reserve (MFR) and quantitative plaque composition | As soon as all required data is available but not later than study completion, an avarage of one year.
  Correlation of MFR on vessel level, expressed as the ratio of Stress/Rest Myocardial Blood Flow (sMBF/rMBF) and plaque composition. Plaque components are defined based on the following Hounsfield Unit (HU) threshold ranges: Low-attenuation plaque: - 100 to 30 HU; Non-calcified plaque: 30 to 350 HU; Calcified plaque: above 350 HU.
Predictive Value of Summed Stress Score (SSS) to lumen stenosis extent on coronary CTA. | As soon as all required data is available but not later than study completion, an avarage of one year.
  The predictive value of semi-quantitative SSS derived from static MPI SPECT using a dedicated software on vessel and participant level to lumen stenosis extent. Classification of SSS is as follows: 0-3 normal, 4-8 mildly abnormal, 8-13 moderately abnormal, and above 13 severely abnormal. The severity of luminal stenosis is defined as follows: no stenosis, 1-24% minimal, 25-49% mild, 50-69% moderate, 70-99% severe, occlusion.
Predictive Value of Summed Stress Score (SSS) to CT-derived Fractional Flow Reserve (FFR-CT) | As soon as all required data is available but not later than study completion, an avarage of one year.
  The predictive value of semi-quantitative SSS derived from static MPI SPECT using a dedicated software on vessel and participant level to FFR-CT of 0.8 or less in any coronary artery. Classification of SSS is as follows: 0-3 normal, 4-8 mildly abnormal, 8-13 moderately abnormal, and above 13 severely abnormal. FFR-CT values are defined as follows: greater than 0.8 is normal, 0.76-0.8 is borderline, and 0.75 or less is abnormal.
Predictive Value of Summed Difference Score (SDS) to lumen stenosis extent on coronary CTA. | As soon as all required data is available but not later than study completion, an avarage of one year.
  The predictive value of semi-quantitative SDS derived from static MPI SPECT using a dedicated software on vessel and participant level to lumen stenosis extent. of 50% or more in the left main coronary artery or 70% or more in any coronary artery. Classification of SDS is as follows: 0-3 normal, 4-8 mildly abnormal, 8-13 moderately abnormal, and above 13 severely abnormal. The severity of luminal stenosis is defined as follows: no stenosis, 1-24% minimal, 25-49% mild, 50-69% moderate, 70-99% severe, occlusion.
Predictive Value of Summed Difference Score (SDS) to CT-derived Fractional Flow Reserve (FFR-CT) | As soon as all required data is available but not later than study completion, an avarage of one year.
  The predictive value of semi-quantitative SDS derived from static MPI SPECT using a dedicated software on vessel and participant level to FFR-CT of 0.8 or less in any coronary artery. Classification of SDS is as follows: 0-3 normal, 4-8 mildly abnormal, 8-13 moderately abnormal, and above 13 severely abnormal. FFR-CT values are defined as follows: greater than 0.8 is normal, 0.76-0.8 is borderline, and 0.75 or less is abnormal.
Comparison of visual assessment of static MPI SPECT to luminal stenosis extent on coronary CTA. | As soon as all required data is available but not later than study completion, an avarage of one year.
  Static MPI SPECT images will be evaluated by a nuclear medicine specialist. Results will be compared to luminal stenosis extent on coronary CTA. The severity of luminal stenosis is defined as follows: no stenosis, 1-24% minimal, 25-49% mild, 50-69% moderate, 70-99% severe, occlusion.
Comparison of visual assessment of static MPI SPECT to CT-derived Fractional Flow Reserve (FFR-CT) | As soon as all required data is available but not later than study completion, an avarage of one year.
  Static MPI SPECT images will be evaluated by a nuclear medicine specialist. Results will be compared to FFR-CT. FFR-CT values are defined as follows: greater than 0.8 is normal, 0.76-0.8 is borderline, and 0.75 or less is abnormal.
Predictive Models of Myocardial Flow Reserve (MFR) and Other Covariants to Coronary Artery Disease (CAD) Severity Identified by Coronary CTA | As soon as all required data is available but not later than study completion, an avarage of one year.
  Composite endpoint:
  model 1: type of chest pain, sex, age model 2: model 1 + static MPI SPECT (SSS, SRS, SDS with the following classification: 0-3 normal, 4-8 mildly abnormal, 8-13 moderately abnormal, and above 13 severely abnormal) model 3: model 2 + MFR (expressed as a sMBF/rMBF ratio) model 4: model 3 + CACS (The following classification is used for CACS: 0, 1-9, 10-99, 100-399, 400-1000, >1000)
Predictive Value of Myocardial Flow Reserve (MFR) to stenosis extent on coronary CTA. | As soon as all required data is available but not later than study completion, an avarage of one year.
  Predictive value of MFR on vessel and participant level, expressed as the ratio of Stress/Rest Myocardial Blood Flow (sMBF/rMBF) to luminal stenosis extent. The severity of luminal stenosis is defined as follows: no stenosis, 1-24% minimal, 25-49% mild, 50-69% moderate, 70-99% severe, occlusion.

CONTACTS AND LOCATIONS:
Overall Officials: Pál Maurovich-Horvat, Prof. Dr., Principal Investigator — Semmelweis University Medical Imaging Centre; Tamás Györke, MD, Study Chair — Semmelweis University Department of Nuclear Medicine
Locations (1):
- Semmelweis University, Medical Imaging Centre, Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
A secure platform will be used to share clinical and imaging data after the results are published.
Time Frame: Clinical and imaging data will be available after the results have been published.
Access Criteria: Access request needs to be made directly to the PI.